CLINICAL TRIAL: NCT04349709
Title: Emotional Dysregulation in Adolescents: Clinical and Biological Correlates.
Brief Title: Emotional Regulation in Teens: Improvement of Constructive Skills
Acronym: EmoTIConS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Responsible Party: Principal Investigator, Laura Pedrini, Principal Investigator, IRCCS Centro San Giovanni di Dio Fatebenefratelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GR-2018-12366754
Record Dates: First submitted 2020-04-10; First posted 2020-04-16 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Emotional Dysregulation
Keywords: Adolescence; Dialectical behavior therapy; stress; school-based intervention; psychoeducation; cortisol; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief school-based DBT-A (Experimental): The students of classes randomized to experimental group receive the brief school-based DBT-A..
  Interventions: Behavioral: Brief school-based DBT-A
- control group (No Intervention): The students of classes randomized to control group continue their school activity as routine.

INTERVENTIONS:
Behavioral: Brief school-based DBT-A — The intervention is inspired to Dialectical Behavior Therapy for Adolescents (DBT-A) (Rathus & Miller, 2015, Mazza et al, 2016; Cappelluccio, 2019). It consists in four monthly 2-hour sessions (for a total of 8 hours) scheduled during school-time. All the sessions are conducted by two psychotherapists trained about DBT. During the sessions, the model of emotions is described through a role-play between conductors. Subsequently, teens are trained about main emotional regulation skills. Moreover, basic elements of distress tolerance, mindfulness and interpersonal efficacy are introduced too.
  Arms: Brief school-based DBT-A

SUMMARY:
This is a prospective randomized study with twofold aim. The first aim is to evaluate the impact of a school-based intervention focused on emotional regulation skills according to Dialectical Behavior Therapy for Adolescents. To this purpose, a sample of students attending the third year of high school (10th grade; 16-19 years) will be recruited, and the interventions will be delivered to the class of students during school-time. The outcomes will be evaluated (post-intervention, 3 and 6-months follow-up) in term of frequency of dysfunctional behaviours, use of emotional regulation skills, and psychological wellbeing. The study is also aimed to identify clinical and biological markers associated to ED in adolescents. To this purpose, youth psychiatric outpatients (16-19 years) will be recruited and compared to the participants of the community sample. All the participants will be evaluated through a comprehensive assessment including both clinical variables and biological variables. Biological evaluations will be conducted to measure cortisol levels during the day (awakening, noon and evening) and the inflammatory profiles

DETAILED DESCRIPTION:
Emotional dysregulation (ED) is a multidimensional construct including lack of awareness and clarity about experienced emotions, nonacceptance of emotional distress, impulsivity, inability to pursue goals when emotionally distressed, and lack of regulatory strategies (Gratz and Roemer, 2004).

The background of the present study is threefold:

1. Adolescence is a heightened risk period for the onset of a wide range of mental disorder. Targeting emotional dysregulation (ED) in adolescence could be particularly relevant, indeed, there is a strong association between ED and dysfunctional behaviours such as substance-related problems (Barahmand et al., 2016; Simons et al., 2017), suicidal ideation (Miller et al., 2017; Rajappa et al., 2012), and self-harm behaviors (Peh et al., 2017).
2. Emotion regulation is a modifiable skill, and school-based prevention programs could be effective for the development of socio-emotional skills, and the improvement of psychological well-being (Taylor et al., 2017).
3. Stressful experiences, especially those occurring early in life, enhance the vulnerability for a spectrum of psychiatric disorders, via targeting both the Hypothalamic-Pituitary-Adrenal (HPA) axis system and the immune/inflammatory system (Lopizzo et al., 2015; 2017). Moreover, there is evidence that individuals exposed to early traumatic experiences exhibit difficulties in regulating their emotional responses (Jennissen et al., 2016). For this reasons, longitudinal studies focused on the association between HPA axis activity and the later development of psychopathology are of great interest because they may be helpful to identify possible risk factors for mental illness. However, only few studies analyzed the neurobiological correlated of ED in adolescents (Goodyer et al., 2000; Halligan et al., 2007).

The main aim of the present study aims to evaluate the impact of an intervention based on Dialectical Behavior Therapy for Adolescents (DBT-A) (Rathus & Miller, 2015, Mazza, et al, 2016) that will be delivered to the class of students during school-time. A total of 426 students attending the third year of high school (10th grade; 16-19 years) will be recruited. In order to optimize the representativeness of the sample, different type of school (i.e. professional institute; technical institute; arts, scientific and classical high schools) will be invited to participate to the study. Moreover, the randomization will be carried out in each school in order to control potential confounding variables associated to a specific type of school. Outcome will be assessed post-intervention, 3 and 6-month follow-up.

The second aim of the present study is to identify clinical and biological markers associated to ED. To this purpose, a clinical sample of youth outpatients (16-19 years) with mental disorders will be recruited and will be compared to the students of the community sample. All the participants will be evaluated through a comprehensive assessment including both clinical variables and biological variables. Clinical assessment will cover different domains: sociodemographic data, emotional dysregulation, psychopathological symptoms, social functioning, childhood trauma, stressful life events during previous year. Biological evaluations will be conducted to measure cortisol levels during the day (awakening, noon and evening) and the inflammatory profiles. Data about biological parameters will permit to investigate whether alterations in biological features related to stress response and inflammation can underlie ED and the vulnerability for psychopathology. Moreover, the same set of biomarkers will be evaluated at the end of the intervention in order to evaluate whether clinical improvements can occur via le modulation of these pathways.

ELIGIBILITY:
Inclusion Criteria:

* Students attending the third year of high school (10th academic grade)
* Signed consent form

Exclusion Criteria:

* Mental retardation
* Asperger syndrome
* Autism spectrum disorders

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 462 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in dysfunctional/impulsive behaviours measured by Checklist for dysfunctional, impulsive behaviours. | 5, 8, 11 months
  The Checklist for dysfunctional, impulsive behaviors is an had-hoc created instrument to measure the dysfunctional/impulsive behaviours (e.g. binge drinking, substance use, unprotected sex, self-harm, etc). For each behaviour, participants are asked to fill the frequency of dysfunctional/impulsive over the previous month
Change in emotional regulation skills measured by the DBT-Ways of Coping Checklist (DBT-WCCL). | 5, 8, 11 months
  The DBT-WCCL is a 59-item self-report instrument measuring the frequency of DBT skills use (DBT Skills Subscale, 38 items) and dysfunctional non-DBT coping strategies (Dysfunctional Coping Subscale, 21 items) over the previous month.

SECONDARY OUTCOMES:
Change in problem-solving strategies as detected by change in mean scores on Social Problem-Solving Inventory-Revised Short Form (SPSI-R:SF) (Maydeu-Olivares & D'Zurilla 1996) | 5, 8, 11 months
  The SPSI-R:SF is a 25-item self-report questionnaire, with five subscales that assess functional and dysfunctional cognitive and emotional orientations towards solving life problems. The subscales are: positive problem orientation (PPO), negative problem orientation (NPO), rational problem solving (RPS), impulsivity-carelessness style (ICS), avoidant style (AS). Higher scores on the NPO, ICS and AS reflect a more maladaptive approach to problem solving; whereas higher scores on the PPO and RPS indicate more adaptive problem solving (D'Zurilla et al., 2002).
Change in depressive symptoms as detected by change in mean Patient Health Questionnaire PHQ-9 global score. | 5, 8, 11 months
  The PHQ is a 9-item self-report questionnaire that cover depressive symptoms criteria of the 9 DSM-IV. A global score is computed as the sum of the nine item and it can range from 0 to 27. Different level of severity of depression can be distinguished according to cut-off (Kroenke et al., 2001).
Change in emotional dysregulation as detected by change in mean scores on the Difficulties in Emotion Regulation Scale (DERS) (Gratz and Roemer, 2004). | 5, 8, 11 months
  The DERS is a 36-item self-report questionnaire with six subscales that assess dimensions of emotional dysregulation: (1) Non-acceptance of emotional responses (6 items); (2) Difficulties engaging in goal-directed behaviour (5 items); (3) Impulse control difficulties (6 items); (4) Lack of emotional awareness (6 items); (5) Limited access to emotion regulation strategies (8 items); (6) Lack of emotional clarity (5 items).

CONTACTS AND LOCATIONS:
Overall Officials: Laura Pedrini, PhD, Principal Investigator — IRCCS Istituto Centro San Giovanni di Dio Fatebenefratelli, Brescia, Italy
Locations (1):
- IRCCS Istituto Centro San Giovanni di Dio Fatebenefratelli, Brescia, Italy

REFERENCES:
- [Background] Mazza et al, DBT Skills in Schools (DBT STEPS-A). Guilford Publications; 2016
- [Background] Rathus&Miller, DBT Skills Manual for Adolescents, Guildford Press; 2015
- [Background] Taylor RD, Oberle E, Durlak JA, Weissberg RP. Promoting Positive Youth Development Through School-Based Social and Emotional Learning Interventions: A Meta-Analysis of Follow-Up Effects. Child Dev. 2017 Jul;88(4):1156-1171. doi: 10.1111/cdev.12864. PMID 28685826
- [Background] Beauchaine TP. Future Directions in Emotion Dysregulation and Youth Psychopathology. J Clin Child Adolesc Psychol. 2015;44(5):875-96. doi: 10.1080/15374416.2015.1038827. Epub 2015 May 27. PMID 26016727
- [Derived] Pedrini L, Rossi R, Magni LR, Lanfredi M, Meloni S, Ferrari C, Macis A, Lopizzo N, Zonca V, Cattaneo A. Emotional Regulation in Teens and Improvement of Constructive Skills (EmoTIConS): study protocol for a randomized controlled trial. Trials. 2021 Dec 14;22(1):920. doi: 10.1186/s13063-021-05886-2. PMID 34906222